CLINICAL TRIAL: NCT01946282
Title: Evidence-Based Colorectal Cancer Screening for the Uninsured
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: PP120229 (IRB# 082012-086)
Record Dates: First submitted 2013-09-13; First posted 2013-09-19 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Colorectal Cancer
Keywords: neoplasm; colorectal; cancer; uninsured; FIT; Fecal Immunochemical Test
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- FIT Invitation Only (Active Comparator): Fecal Immunochemical Test (FIT) mailed to patient homes free of charge.
  Intervention: Fecal Immunochemical Test (FIT) kits and an invitation letter to complete colorectal cancer screening are mailed to the homes of study eligible patients. A postage paid return mailer is included. Automated and "live" phone call reminders are made at the time of invitation and within one week of invitation. Up to two "live" phone call reminders are attempted 2 to 3 weeks post invitation.
  Follow up for patients who return a normal test in Year 1 will consist of repeat screening invitations in Year 2 and Year 3 consistent with guideline recommended annual FIT for colorectal cancer screening. Follow up for patients who return an abnormal test will consist of navigation to complete colonoscopy.
  Interventions: Other: FIT Invitation Only
- FIT plus $5 Incentive (Active Comparator): Fecal Immunochemical Test (FIT) mailed to patient homes, plus an incentive to complete the test.
  Intervention: FIT kits and invitation letter with a $5 gift card incentive to complete screening are mailed to the homes of 1000 randomly assigned eligible patients. A postage paid return mailer is included. Automated and "live" phone call reminders are made at the time of invitation and within one week of invitation. Up to two "live" phone call reminders are attempted 2 to 3 weeks post invitation.
  Follow up for patients who return a normal test in Year 1 will consist of repeat screening invitations in Year 2 and Year 3. Follow up for patients who return an abnormal test will consist of navigation to complete colonoscopy.
  Interventions: Other: FIT plus $5 Incentive
- FIT plus $10 Incentive (Active Comparator): Fecal Immunochemical Test (FIT) mailed to patient homes, plus an incentive to complete the test.
  Intervention: FIT kits and invitation letter with a $10 gift card incentive to complete screening are mailed to the homes of 1000 randomly assigned eligible patients. A postage paid return mailer is included. Automated and "live" phone call reminders are made at the time of invitation and within one week of invitation. Up to two "live" phone call reminders are attempted 2 to 3 weeks post invitation.
  Follow up for patients who return a normal test in Year 1 will consist of repeat screening invitations in Year 2 and Year 3. Follow up for patients who return an abnormal test will consist of navigation to complete colonoscopy.
  Interventions: Other: FIT plus $10 Incentive

INTERVENTIONS:
Other: FIT Invitation Only — Patients meeting the inclusion / exclusion criteria are mailed invitations to complete a free colorectal cancer screening. POLYMEDCO Fecal Immunochemical Tests (FIT) are mailed to patient homes with instructions, followed up with live and TELEVOX reminder phone calls.
  Other Names: POLYMEDCO Fecal Immunochemical Test (FIT); John Peter Smith Health System
  Arms: FIT Invitation Only
Other: FIT plus $5 Incentive — Patients meeting the inclusion / exclusion criteria are mailed invitations to complete a free colorectal cancer screening. POLYMEDCO Fecal Immunochemical Tests (FIT) are mailed to patient homes with instructions, followed up with live and TELEVOX reminder phone calls. Patients are offered a small incentive to complete their screening.
  Other Names: POLYMEDCO Fecal Immunochemical Test (FIT); John Peter Smith Health System
  Arms: FIT plus $5 Incentive
Other: FIT plus $10 Incentive — Patients meeting the inclusion / exclusion criteria are mailed invitations to complete a free colorectal cancer screening. POLYMEDCO Fecal Immunochemical Tests (FIT) are mailed to patient homes with instructions, followed up with live and TELEVOX reminder phone calls. Patients are offered a small incentive to complete their screening.
  Other Names: POLYMEDCO Fecal Immunochemical Test (FIT)
  Arms: FIT plus $10 Incentive

SUMMARY:
Through this program, the investigators will test a systematic colon cancer screening outreach strategy for increasing screening completion among uninsured patients, not up-to-date with screening. The intervention will consist of mailed screening invitations, with processes such as phone reminders to promote screening and evidence based follow up. All patients will be randomly assigned to receive mailed invitations to complete a home fecal immunochemical test (FIT). Some patients will be randomly assigned to receive a small financial incentive on completion of FIT testing.

DETAILED DESCRIPTION:
All patients meeting inclusion/exclusion criteria will receive mailed invitation and FIT kit to complete screening, with processes to promote screening completion. The list of eligible patients will be divided into 5 groups so that the expected group of 10,000 patients will receive invitations spread out in time, so as to avoid overwhelming the system. The invitation letters emphasize importance of colorectal cancer screening, encourage the patient to complete FIT screening with the enclosed FIT kit, and will be signed by John Pter Smith (JPS) investigators as representatives of JPS primary care physicians.

The invitation kit will include a 1-sample POLYMEDCO Sensor FIT, including simplified instructions on how to perform the test, as well as a return mailer with prepaid postage. Diet/medication restriction will not be required. Kits will be returned to JPS and processed per manufacturer recommendations.

Automated and "live" phone call reminders to encourage screening completion will be sent at time of invite and within week 1 of the invitation. Up to two "live" phone call reminders will be attempted 2 to 3 weeks post invitation, using English and Spanish standard scripts.

Follow up for patients with a normal test in Year 1 will consist of repeat screening invitations in Year 2 and Year 3 consistent with guideline recommended annual FIT for colorectal screening. Follow up for patients with an abnormal FIT will consist of navigation to complete a colonoscopy. Patients with abnormal FIT will be called by the screening team within 1 week to report the result and facilitate direct scheduling of colonoscopy or a pre-colonoscopy visit. Follow up of patients with a colorectal cancer will consist of navigation to first treatment consultation visit. A surgery or oncology clinic follow up will be scheduled for all patients with a colorectal cancer diagnosis if such follow up is not already scheduled by the colonoscopist who diagnosed the colorectal cancer. Reminder calls for these visits will be made daily for up to one week.

A group of 2,000 individuals will be randomly assigned to receive a modest financial incentive to complete screening, in addition to the organized outreach program. The incentive will consist of a gift card in one of two small dollar amounts to a local retailer. Incentives will be mailed by the JPS outreach team, in exchange for successful FIT completion, after the FIT has been returned.

Follow up for determining screening completion for all included patients will be through the end of Year 3 regardless of whether or not patients respond to screening invitations. Once included, patients will remain in the program unless they no longer meet age criteria. Patients in both the standard (non-incentive) and incentive invitation groups who do not respond to initial invitation will be followed for screening outcomes, but will not receive repeat invitations. For patients who die on follow up or who do not have additional health system encounters, follow up will be censored at time of death or last health encounter, respectively.

Each year, patients who newly meet our inclusion/exclusion criteria will be included in the program. For example, patients newly turning 50 in year 2 or 3 meeting all other inclusion/exclusion criteria will receive screening outreach. Similarly, a 60 year old patient new to the JPS system and meeting inclusion/exclusion criteria will also receive screening outreach.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-64.
* Uninsured, but participants in John Peter Smith Health System (JPS) medical assistance program for the uninsured.
* One or more visits to a JPS primary care clinic within a year.
* Not up-to-date with colorectal cancer screening.

Exclusion Criteria:

* Patients with a history of Colorectal Cancer or colon resection, no address and/or phone number on file, or who are incarcerated will be excluded.

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8565 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Argenbright, M.D., Principal Investigator — University of Texas Southwestern Medical Center; Samir Gupta, M.D., Study Director — University of California, San Diego

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Siegel R, Xu J, Ward E. Cancer statistics, 2010. CA Cancer J Clin. 2010 Sep-Oct;60(5):277-300. doi: 10.3322/caac.20073. Epub 2010 Jul 7. PMID 20610543
- [Background] StatBite: National Costs for Cancer Care in 2010 in Billions of Dollars by Cancer Site. J Natl Cancer Inst. 2012 Jan 4;104(1):13. doi: 10.1093/jnci/djr534. Epub 2011 Dec 14. No abstract available. PMID 22173584
- [Background] Ward E, Halpern M, Schrag N, Cokkinides V, DeSantis C, Bandi P, Siegel R, Stewart A, Jemal A. Association of insurance with cancer care utilization and outcomes. CA Cancer J Clin. 2008 Jan-Feb;58(1):9-31. doi: 10.3322/CA.2007.0011. Epub 2007 Dec 20. PMID 18096863
- [Background] Hardcastle JD, Chamberlain JO, Robinson MH, Moss SM, Amar SS, Balfour TW, James PD, Mangham CM. Randomised controlled trial of faecal-occult-blood screening for colorectal cancer. Lancet. 1996 Nov 30;348(9040):1472-7. doi: 10.1016/S0140-6736(96)03386-7. PMID 8942775
- [Background] Mandel JS, Bond JH, Church TR, Snover DC, Bradley GM, Schuman LM, Ederer F. Reducing mortality from colorectal cancer by screening for fecal occult blood. Minnesota Colon Cancer Control Study. N Engl J Med. 1993 May 13;328(19):1365-71. doi: 10.1056/NEJM199305133281901. PMID 8474513
- [Background] Kronborg O, Fenger C, Olsen J, Jorgensen OD, Sondergaard O. Randomised study of screening for colorectal cancer with faecal-occult-blood test. Lancet. 1996 Nov 30;348(9040):1467-71. doi: 10.1016/S0140-6736(96)03430-7. PMID 8942774
- [Background] Faivre J, Dancourt V, Lejeune C, Tazi MA, Lamour J, Gerard D, Dassonville F, Bonithon-Kopp C. Reduction in colorectal cancer mortality by fecal occult blood screening in a French controlled study. Gastroenterology. 2004 Jun;126(7):1674-80. doi: 10.1053/j.gastro.2004.02.018. PMID 15188160
- [Background] Atkin WS, Edwards R, Kralj-Hans I, Wooldrage K, Hart AR, Northover JM, Parkin DM, Wardle J, Duffy SW, Cuzick J; UK Flexible Sigmoidoscopy Trial Investigators. Once-only flexible sigmoidoscopy screening in prevention of colorectal cancer: a multicentre randomised controlled trial. Lancet. 2010 May 8;375(9726):1624-33. doi: 10.1016/S0140-6736(10)60551-X. Epub 2010 Apr 27. PMID 20430429
- [Background] Kahi CJ, Imperiale TF, Juliar BE, Rex DK. Effect of screening colonoscopy on colorectal cancer incidence and mortality. Clin Gastroenterol Hepatol. 2009 Jul;7(7):770-5; quiz 711. doi: 10.1016/j.cgh.2008.12.030. Epub 2009 Jan 11. PMID 19268269
- [Background] Brenner H, Chang-Claude J, Seiler CM, Rickert A, Hoffmeister M. Protection from colorectal cancer after colonoscopy: a population-based, case-control study. Ann Intern Med. 2011 Jan 4;154(1):22-30. doi: 10.7326/0003-4819-154-1-201101040-00004. PMID 21200035
- [Background] Baxter NN, Goldwasser MA, Paszat LF, Saskin R, Urbach DR, Rabeneck L. Association of colonoscopy and death from colorectal cancer. Ann Intern Med. 2009 Jan 6;150(1):1-8. doi: 10.7326/0003-4819-150-1-200901060-00306. Epub 2008 Dec 15. PMID 19075198
- [Derived] Jetelina KK, Yudkin JS, Miller S, Berry E, Lieberman A, Gupta S, Balasubramanian BA. Patient-Reported Barriers to Completing a Diagnostic Colonoscopy Following Abnormal Fecal Immunochemical Test Among Uninsured Patients. J Gen Intern Med. 2019 Sep;34(9):1730-1736. doi: 10.1007/s11606-019-05117-0. Epub 2019 Jun 21. PMID 31228053
- [Derived] Berry E, Miller S, Koch M, Balasubramanian B, Argenbright K, Gupta S. Lower Abnormal Fecal Immunochemical Test Cut-Off Values Improve Detection of Colorectal Cancer in System-Level Screens. Clin Gastroenterol Hepatol. 2020 Mar;18(3):647-653. doi: 10.1016/j.cgh.2019.04.077. Epub 2019 May 11. PMID 31085338

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18,700 age-eligible patients with qualifying outpatient clinic visits were identified for invitation. 10,135 patients were excluded from participation due to the following: primary language not English or Spanish, missing contact information, incarceration, screen up-to-date, and prior history of colorectal cancer or inflammatory bowel disease.
Groups:
- FIT Invitation Only, No Incentive: Fecal Immunochemical Test (FIT) mailed to patient homes free of charge. Fecal Immunochemical Test (FIT) kits and an invitation letter to complete colorectal cancer screening are mailed to the homes of study eligible patients. A postage paid return mailer is included. Automated and "live" phone call reminders are made at the time of invitation and within 1 week of invitation. Up to two "live" phone call reminders are attempted 2 to 3 weeks post invitation.
  Follow up for patients who return a normal test in Year 1 will consist of repeat screening invitations in Year 2 and Year 3 consistent with guideline recommended annual FIT for colorectal cancer screening. Follow up for patients who return an abnormal test will consist of navigation to complete colonoscopy.
- FIT Plus $5 Incentive: Fecal Immunochemical Test (FIT) mailed to patient homes, plus an $5 gift card incentive to complete the test. FIT kits and invitation letter with a gift card incentive to complete screening are mailed to the homes of 1000 randomly assigned eligible patients. A postage paid return mailer is included. Automated and "live" phone call reminders are made at the time of invitation and within 1 week of invitation. Up to two "live" phone call reminders are attempted 2 to 3 weeks post invitation.
  Follow up for patients who return a normal test in Year 1 will consist of repeat screening invitations in Year 2 and Year 3. Follow up for patients who return an abnormal test will consist of navigation to complete colonoscopy.
- FIT Plus $10 Incentive: Fecal Immunochemical Test (FIT) mailed to patient homes, plus an $10 gift card incentive to complete the test. FIT kits and invitation letter with a gift card incentive to complete screening are mailed to the homes of 1000 randomly assigned eligible patients. A postage paid return mailer is included. Automated and "live" phone call reminders are made at the time of invitation and within 1 week of invitation. Up to two "live" phone call reminders are attempted 2 to 3 weeks post invitation.
  Follow up for patients who return a normal test in Year 1 will consist of repeat screening invitations in Year 2 and Year 3. Follow up for patients who return an abnormal test will consist of navigation to complete colonoscopy.
Period: Year 1
Arm/Group | FIT Invitation Only, No Incentive | FIT Plus $5 Incentive | FIT Plus $10 Incentive
Started | 6565 | 1000 | 1000
Completed (Number of returned FIT kits) | 2379 | 392 | 346
Not Completed | 4186 | 608 | 654
Not completed — Did not return FIT kit | 4186 | 608 | 654
Period: Year 2
Arm/Group | FIT Invitation Only, No Incentive | FIT Plus $5 Incentive | FIT Plus $10 Incentive
Started | 2051 (Patients are those with Year 1 negative FIT results, or no longer met inclusion criteria.) | 341 (Patients are those with Year 1 negative FIT results, or no longer met inclusion criteria.) | 299 (Patients are those with Year 1 negative FIT results, or no longer met inclusion criteria.)
Completed | 1248 | 210 | 184
Not Completed | 803 | 131 | 115
Not completed — Did not return FIT kit | 803 | 131 | 115
Period: Year 3
Arm/Group | FIT Invitation Only, No Incentive | FIT Plus $5 Incentive | FIT Plus $10 Incentive
Started | 1144 (Patients are those with Year 2 negative FIT results, or no longer met inclusion criteria.) | 184 (Patients are those with Year 2 negative FIT results, or no longer met inclusion criteria.) | 170 (Patients are those with Year 2 negative FIT results, or no longer met inclusion criteria.)
Completed | 856 | 141 | 140
Not Completed | 288 | 43 | 30
Not completed — Did not return FIT kit | 288 | 43 | 30

BASELINE CHARACTERISTICS:
Population: Baseline participants meeting inclusion criteria were randomized and invited in Year 1.
Groups:
- FIT Invitation Only: Fecal Immunochemical Test (FIT) mailed to patient homes free of charge. Fecal Immunochemical Test (FIT) kits and an invitation letter to complete colorectal cancer screening are mailed to the homes of study eligible patients. A postage paid return mailer is included. Automated and "live" phone call reminders are made at the time of invitation and within one week of invitation. Up to two "live" phone call reminders are attempted 2 to 3 weeks post invitation.
  Follow up for patients who return a normal test in Year 1 will consist of repeat screening invitations in Year 2 and Year 3 consistent with guideline recommended annual FIT for colorectal cancer screening. Follow up for patients who return an abnormal test will consist of navigation to complete colonoscopy.
  FIT Invitation Only: Patients meeting the inclusion / exclusion criteria are mailed invitations to complete a free colorectal cancer screening. POLYMEDCO Fecal Immunochemical Tests (FIT) are mailed to patient homes.
- FIT Plus $5 Incentive; FIT Plus $10 Incentive: Fecal Immunochemical Test (FIT) mailed to patient homes, plus an incentive to complete the test. FIT kits and invitation letter with a gift card incentive in one of two small dollar amounts to complete screening are mailed to the homes of 2000 (1000 per group) randomly assigned eligible patients. A postage paid return mailer is included. Automated and "live" phone call reminders are made at the time of invitation and within one week of invitation. Up to two "live" phone call reminders are attempted 2 to 3 weeks post invitation.
  Follow up for patients who return a normal test in Year 1 will consist of repeat screening invitations in Year 2 and Year 3. Follow up for patients who return an abnormal test will consist of navigation to complete colonoscopy.
  FIT plus Incentive: Patients meeting the inclusion / exclusion criteria are mailed invitations to complete a free colorectal cancer screening. POLYMEDCO Fecal Immunochemical Tests (FIT) are mailed to patient homes.
- Total: Total of all reporting groups
Arm/Group | FIT Invitation Only | FIT Plus $5 Incentive | FIT Plus $10 Incentive | Total
Number analyzed (Participants) | 6565 | 1000 | 1000 | 8565
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [53 to 60] | 56 [53 to 60] | 56 [53 to 60] | 56 [53 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4042 | 610 | 644 | 5296
  Male | 2523 | 390 | 356 | 3269
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2428 | 381 | 368 | 3177
  Black | 1578 | 270 | 245 | 2093
  Hispanic | 1951 | 257 | 293 | 2501
  Asian | 127 | 19 | 23 | 169
  Other | 405 | 59 | 54 | 518
  Unknown | 76 | 14 | 17 | 107

OUTCOME MEASURES:

1. Primary Outcome: FIT Completion Among Patients Offered Any Incentive vs. Outreach Alone Each Year
Description: Primary outcome was analyzed using an intent-to-screen approach where a 2-sided P-value <0.05 was considered statistically significant. Patients were randomly assigned to one of 3 groups: outreach only, outreach + $5 incentive upon FIT return, and outreach + $10 incentive upon FIT return. For analysis, incentive groups were combined and compared to outreach alone.
Time Frame: Each year for three years
Population: If FIT is positive, patients are routed to appropriate treatment. If FIT is negative, patients mailed invitations in the following year.
Measure: Count of Participants; unit: Participants
Groups:
- Standard Invite: Fecal Immunochemical Test (FIT) kits and an invitation letter to complete colorectal cancer screening are mailed to the homes of study eligible patients. A postage paid return mailer is included. Automated and "live" phone call reminders are made at the time of invitation and within one week of invitation. Up to two "live" phone call reminders are attempted 2 to 3 weeks post invitation.
- Incentive Invite: The denominator population for evaluating baseline and end of Year 3 screening rates will consist of patients meeting the following criteria: 1) Age 50-64, 2) Uninsured, but participants in JPS's medical assistance program for the uninsured, 3) One or more visits to a JPS primary care clinic within a year, 4) Address and phone number on file, 5) No history of CRC or colon resection, 6) Not incarcerated
Arm/Group | Standard Invite | Incentive Invite
Number analyzed (Participants) | 6565 | 2000
Participants
  Year 1 Screening Rate | 2391 | 738
  Year 2 Screening Rate: number analyzed (Participants) | 2051 | 640
  Year 2 Screening Rate | 1255 | 394
  Year 3 Screening Rate: number analyzed (Participants) | 1144 | 354
  Year 3 Screening Rate | 856 | 281
Statistical Analysis 1: Comparison: Standard Invite vs Incentive Invite; Test type: Equivalence — Assuming a FIT return rate of 29% for the outreach only group at an a=0.05, we estimated more than 90% power to detect an absolute difference greater than 5% when using a chi-square test of proportions to compare patients who received any incentive ($5 or $10) compared with patients who received outreach only; p = 0.59, Chi-squared
Statistical Analysis 2: Comparison: Standard Invite vs Incentive Invite; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .75, Chi-squared
Statistical Analysis 3: Comparison: Standard Invite vs Incentive Invite; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = .080, Chi-squared

2. Secondary Outcome: FIT Completion for Groups Offered $5 vs. Outreach Alone, $10 vs. Outreach Alone, and $5 vs. $10 Incentive
Description: Patients were randomly assigned to one of 3 groups: outreach only, outreach + $5 incentive upon FIT return, and outreach + $10 incentive upon FIT return. In year 4, use of financial incentives were discontinued and all patients with a normal result in year 3 were invited to complete a FIT using outreach only, regardless of their original intervention group.
Time Frame: Each year for three years
Population: Patients were re-invited after participation in previous year and had a negative FIT result.
Measure: Count of Participants; unit: Participants
Groups:
- $5 Incentive Invitation: Fecal Immunochemical Test (FIT) mailed to patient homes free of charge. Fecal Immunochemical Test (FIT) kits and an invitation letter to complete colorectal cancer screening are mailed to the homes of study eligible patients. A postage paid return mailer is included. Automated and "live" phone call reminders are made at the time of invitation and within one week of invitation. Up to two "live" phone call reminders are attempted 2 to 3 weeks post invitation.
  Follow up for patients who return a normal test in Year 1 will consist of repeat screening invitations in Year 2 and Year 3 consistent with guideline recommended annual FIT for colorectal cancer screening. Follow up for patients who return an abnormal test will consist of navigation to complete colonoscopy.
- $10 Incentive Invite: Fecal Immunochemical Test (FIT) mailed to patient homes, plus an incentive to complete the test. FIT kits and invitation letter with a gift card incentive in one of two small dollar amounts to complete screening are mailed to the homes of 2000 (1000 per group) randomly assigned eligible patients. A postage paid return mailer is included. Automated and "live" phone call reminders are made at the time of invitation and within one week of invitation. Up to two "live" phone call reminders are attempted 2 to 3 weeks post invitation.
  Follow up for patients who return a normal test in Year 1 will consist of repeat screening invitations in Year 2 and Year 3. Follow up for patients who return an abnormal test will consist of navigation to complete colonoscopy.
  FIT plus Incentive: Patients meeting the inclusion / exclusion criteria are mailed invitations to complete a free colorectal cancer screening. POLYMEDCO Fecal Immunochemical Tests (FIT) are mailed to patient homes.
- Outreach Alone: The outreach included: (i) a mailed invitation to complete and return the FIT in English and Spanish; (ii) a 1-sample Polymedco OC Sensor FIT test; (iii) 2 automated telephone reminders in English and Spanish at the time invitations were mailed and 1 week later, encouraging test completion; and (iv) up to 2 live telephone reminders within 3 weeks of the invitation mailing, if the FIT was not returned or if the patient had not been reached during earlier attempts.
Arm/Group | $5 Incentive Invitation | $10 Incentive Invite | Outreach Alone
Number analyzed (Participants) | 1000 | 1000 | 6565
Participants
  Year 1 Initial Screening Rate | 392 | 346 | 2379
  Year 2 Repeat Screening Rate: number analyzed (Participants) | 341 | 299 | 2051
  Year 2 Repeat Screening Rate | 210 | 184 | 1248
  Year 3 Repeat Screening Rate: number analyzed (Participants) | 184 | 170 | 1144
  Year 3 Repeat Screening Rate | 141 | 140 | 856
Statistical Analysis 1: Comparison: $5 Incentive Invitation vs Outreach Alone; Test type: Equivalence — Based on design, at a significance level of 0.05 group size was set to detect an minimum absolute difference in return rate of 10%, while maintaining more than 90% power. Baseline return rates were projected per group using prior study data: 29% for the outreach only group, 45% in the $5 incentive group, and 53% in the $10 incentive group; p = 0.070, Chi-squared
Statistical Analysis 2: Comparison: $5 Incentive Invitation vs Outreach Alone; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.80, Chi-squared
Statistical Analysis 3: Comparison: $5 Incentive Invitation vs Outreach Alone; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.60, Chi-squared
Statistical Analysis 4: Comparison: $10 Incentive Invite vs Outreach Alone; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.31, Chi-squared
Statistical Analysis 5: Comparison: $10 Incentive Invite vs Outreach Alone; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.82, Chi-squared
Statistical Analysis 6: Comparison: $10 Incentive Invite vs Outreach Alone; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.033, Chi-squared
Statistical Analysis 7: Comparison: $5 Incentive Invitation vs $10 Incentive Invite; Test type: Equivalence — We estimated needing 545 observations per incentive group to achieve power necessary to detect at least a 10% absolute difference in FIT return rate between patients who received the $5 incentive versus patients who received the $10 incentive, with assumed rates of 45% in the $5 incentive group and 53% in the $10 incentive group, a=0.05, and power=90%; p = 0.033, Chi-squared
Statistical Analysis 8: Comparison: $5 Incentive Invitation vs $10 Incentive Invite; Test type: Equivalence; p > 0.99, Chi-squared
Statistical Analysis 9: Comparison: $5 Incentive Invitation vs $10 Incentive Invite; Test type: Equivalence; p = 0.184, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse event data was assessed for each subject starting from study enrollment (initial mailing of study invitation) until the end of patient follow up for each year of participation in the study (through the completion of all applicable screening and/or diagnostic follow up as a result of study invitation). The entire duration of adverse event monitoring is subject dependent upon how long the particular subject participated in the study.
Description: No adverse events were experienced by subjects during this research.
Groups:
- FIT Invitation Only, No Incentive: Fecal Immunochemical Test (FIT) mailed to patient homes free of charge. Fecal Immunochemical Test (FIT) kits and an invitation letter to complete colorectal cancer screening are mailed to the homes of study eligible patients. A postage paid return mailer is included. Automated and "live" phone call reminders are made at the time of invitation and within 1 week of invitation. Up to two "live" phone call reminders are attempted 2 to 3 weeks post invitation.
- FIT Plus $5 Incentive; FIT Plus $10 Incentive: Fecal Immunochemical Test (FIT) mailed to patient homes, plus an incentive to complete the test. FIT kits and invitation letter with a gift card incentive in one of two small dollar amounts to complete screening are mailed to the homes of 2000 (1000 per group) randomly assigned eligible patients. A postage paid return mailer is included. Automated and "live" phone call reminders are made at the time of invitation and within 1 week of invitation. Up to two "live" phone call reminders are attempted 2 to 3 weeks post invitation.
Arm/Group | FIT Invitation Only, No Incentive | FIT Plus $5 Incentive | FIT Plus $10 Incentive
All-Cause Mortality (participants affected / at risk) | 0/6565 | 0/1000 | 0/1000
Serious Adverse Events (participants affected / at risk) | 0/6565 | 0/1000 | 0/1000
Other Adverse Events (participants affected / at risk) | 0/6565 | 0/1000 | 0/1000

LIMITATIONS AND CAVEATS:
We focused exclusively on an uninsured low-income population and offered relatively modest incentives. Thus, our results may not be generalizable to other populations or incentive amounts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT01946282/Prot_SAP_000.pdf